CLINICAL TRIAL: NCT05974488
Title: The Efficacy of Distal Pharyngeal Airway in Enhancing Oxygenation During Transesophageal Echocardiography (TEE) in Patients Sedated With Propofol
Brief Title: The Efficacy of Distal Pharyngeal Airway for Oxygenation During TEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Fouad souki, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20221246
Record Dates: First submitted 2023-05-31; First posted 2023-08-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Distal Pharyngeal Airway (Experimental): Participants in this group will use the McMurray enhanced airway to have oxygen delivered throughout a TEE procedure for up to 60 minutes.
  Interventions: Device: McMurray Enhanced Airway
- Nasal cannula group (Active Comparator): Participant in this group will receive oxygen through a nasal cannula during the TEE procedure for up to 60 minutes.
  Interventions: Device: Nasal Cannula

INTERVENTIONS:
Device: McMurray Enhanced Airway — The MEA is non-sterile. It can be used in inpatient or outpatient surgery, in hospital or clinic settings, or in an emergency setting. The MEA has five parts: an optional 15 mm connector, flange (color-coded for size), elongated cushioned bite block, flexible cannula, and distal tip, and a channel to allow for passage of air and a suction catheter. The MEA is designed to open and maintain a patient's upper airway. Oxygen will be delivered through the breathing circuit with the following parameters: 40% oxygen at 6 liters/min flow throughout the procedure time. The MEA will be placed in the participant's oropharyngeal airway one time during an in-person visit.
  Arms: Distal Pharyngeal Airway
Device: Nasal Cannula — Participants in this group will use the nasal cannula to deliver oxygen as per standard of care one time during the in-person visit.
  Arms: Nasal cannula group

SUMMARY:
The purpose of this study is to investigate the effect of using the McMurray Enhanced Airway (MEA) which is a flexible extended-length distal pharyngeal airway on improving oxygen delivery compared to standard nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients scheduled to undergo an elective TEE procedure.

Exclusion Criteria:

* Patients with history of uncontrolled gastroesophageal reflux disease
* Patients with anatomical airway obstruction
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxia | during procedure (up to 60 minutes)
  Determine the incidence of hypoxia defined as oxygen saturation by pulse oximetry (SPo2)= 75-89%.

SECONDARY OUTCOMES:
Incidence of subclinical hypoxia | during procedure (up to 60 minutes)
  Determine the incidence of subclinical hypoxia defined as SPo2= 90-95%.
Incidence of severe Hypoxia | during procedure (up to 60 minutes)
  Determine the incidence of severe hypoxia defined as SPo2<75%.

CONTACTS AND LOCATIONS:
Overall Officials: Fouad G Souki, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No